CLINICAL TRIAL: NCT02538978
Title: Safety and Effectiveness of the SurgWerksTM-CLI Kit and VXPTM System for the Rapid Intra-operative Aspiration, Preparation and Intramuscular Injection of Concentrated Autologous Bone Marrow Cells Into the Ischemic Index Limb of Rutherford Category 5 Non-Reconstructable Critical Limb Ischemia Patients
Brief Title: Critical Limb Ischemia Rapid Delivery by SurgWerks-CLI Kit and VXP System
Acronym: CLIRST III
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cesca Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CST/CLI/143003
Record Dates: First submitted 2015-08-18; First posted 2015-09-02 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Critical Limb Ischemia (CLI)
Keywords: CLI
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Device Arm (Experimental): Device arm subjects will receive an intra-operative point of care aspiration, preparation and intramuscular injection of autologous bone marrow concentrate (aBMC) into the afflicted lower index limb.
  Interventions: Biological: Autologous Bone Marrow Concentrate (aBMC)
- Placebo Arm (Placebo Comparator): Placebo arm subjects will undergo an intra-operative point of care aspiration and preparation of bone marrow via the investigational device exactly as the Treatment Arm. However, instead of receiving the dosing with the aBMC device output, they will receive an intramuscular injection of diluted autologous peripheral blood into the afflicted lower index limb.
  Interventions: Biological: Placebo Control (diluted autologous peripheral blood)

INTERVENTIONS:
Biological: Autologous Bone Marrow Concentrate (aBMC) — Aspirated bone marrow will be processed by centrifugation, separating out a concentrate (aBMC) comprising primarily white blood cells and platelets. These cells will be injected i.m. to loci determined by the operating physician using imaging and vascular flow criteria.
  Device: SurgWerks-CLI Kit
  Device: VXP System
  Arms: Device Arm
Biological: Placebo Control (diluted autologous peripheral blood) — Diluted peripheral blood prepared in a blinded fashion to resemble bone marrow will be injected intramuscularly per the same procedure used for the Experimental Device Arm.
  Other Names: Diluted autologous peripheral blood
  Arms: Placebo Arm

SUMMARY:
This is a prospective, double-blinded, randomized, placebo-controlled, multi-center, pivotal clinical study in which subjects are evaluated for prevention of major limb amputation in the treatment of non-reconstructable Rutherford Category 5 critical limb ischemia (CLI). Subjects will be randomized in 3:1 ratio (device treatment: placebo-control).

DETAILED DESCRIPTION:
Device arm subjects will receive an intra-operative point of care aspiration, preparation and intramuscular injection of autologous bone marrow cell concentrate (aBMC) into the afflicted lower index limb.

Bone marrow will be collected bilaterally from the patient's iliac crests using the SurgWerks-CLI Kit aspiration trocar under local anesthesia with mild to moderate sedation or general anesthesia, processed through the VXP System device to yield a rich cell and plasma concentrate ("aBMC"). Additionally, 10 mL of autologous peripheral blood will be aspirated for the placebo preparation.

The Treatment Arm will receive the aBMC, which will be intramuscularly injected at multiple mapped sites/angiosomes into the ischemic index limb using the SurgWerks-CLI Kit supplied Therapeutic Infusion Needles and standard hypodermic needles. The procedure will be performed in a surgical suite and will take approximately 1.5-2.0 hours to complete. The subjects will be observed for 24 hours following the procedure for observation and control as necessary of post-operative pain, bleeding, and infection.

Placebo Arm subjects will undergo an intra-operative point of care aspiration and preparation of bone marrow via the investigational device exactly as the Treatment Arm. However, instead of receiving the dosing with the aBMC device output, they will receive an intramuscular injection of diluted autologous peripheral blood into the afflicted lower index limb.

At pre-specified follow-up intervals, all subjects in each arm will be evaluated for:

* Major limb amputation free survival
* Time to Treatment Failure (TTF)
* Wound healing: Quantitative evaluation of wound(s)
* Quality of life assessment (VascuQoL and SF-36)
* Skin Perfusion Pressure (SPP) - Quantitative evaluation of blood flow
* Rest pain assessment
* Brachial Index (ABI)

ELIGIBILITY:
Inclusion Criteria

IC 1 Male or Female of age ≥ 40 and ≤ 85 years.

* IC 2 Chronic CLI from atherosclerotic ischemic peripheral arterial disease (PAD) of a lower limb classified as Rutherford Category 5: (ischemic pain at rest and minor tissue loss with ulceration per IC 3).
* IC 3 Ulcer of the toe(s) and/or foot (below the ankle) having a total tissue loss (full thickness) of at least 0.5 cm2 but no greater than 20 cm2 (0.5 cm2 ≤ wound area ≤ 20 cm2) or greater than 10 cm2 on the heel. Note: exposed tendon or bone is an exclusion, see EC 7
* IC 4 A non-surgical candidate for revascularization as ruled by the investigator and confirmed by the BICR (single reader) and defined as: failure of all previous standard revascularization therapies /reconstruction attempts (at least two weeks prior to enrollment) no conduit suitable for bypass grafting, medical high risk that precludes bypass surgery, and diffuse multi-segment disease, or extensive infra-popliteal disease not amenable to endovascular therapy..
* IC 5 Ability to maintain compliance with tolerated medical management regimen for PAD that includes smoking cessation, and may include management of hyperlipidemia, diabetic management, antiplatelet therapy, statin therapy, ACE inhibitor therapy (or ARB therapy) and beta blocker therapy for control of blood pressure.
* IC 6 Willingness, ability and commitment to participate in baseline and follow-up evaluations for the full length of the study.
* IC 7 Poor lower extremity perfusion defined as an:

  * ABI ≤ 0.6, or
  * Foot/Ankle SPP ≤ 30 mmHg, or
  * Ankle systolic pressure ≤ 60 mmHg or Toe pressure <40 mmHg
* IC 8 Written informed consent.

Exclusion Criteria

* EC1 Women who are pregnant, lactating or planning a pregnancy during the twelve (12) months of the follow-up period.
* EC2 Advanced CLI of the affected index limb classified in a category other than Rutherford 5.
* EC3 Advanced CLI in the opposing limb (non-index) with Rutherford category 6.
* EC4 Patients with aorta-iliac occlusive disease with >50% stenosis
* EC5 Any prior amputation in the index limb beyond the toe(s) or digits or trans-metatarsal in the past four weeks.
* EC6 Ischemic wounds with systemic infectious symptoms (fever, hypotension, and/or positive blood cultures).
* EC7 Ischemic wounds having exposed tendon or bone.
* EC8 PT/INR > 2.0 in the pre-admission baseline. If on warfarin, PT/INR which is not titrated to ≥ 2.0 prior to the treatment procedure.
* EC9 Ulcers above the ankle
* EC10 Subjects on renal dialysis or with end stage renal disease (Serum creatinine of ≥ 2.5 mg/dl or GFR ≤ 15 using CKD-EPI equation of National Kidney Foundation).
* EC11 Poorly controlled diabetes mellitus (HbA1c ≥ 10%)
* EC12 Anemia defined as a Hgb of ≤ 10mg/dl or a HCT ≤ 30%
* EC13 Any diagnosed immune-deficient status except well-controlled HIV infection (defined as HIV RNA qPCR ≤ 20 copies/mL).
* EC14 History of any neoplastic disease/cancer (other than basal cell carcinoma) in the previous three (3) years.
* EC15 Intolerance to heparin.
* EC16 Contraindicated to CT angiography.
* EC17 Medical risk that precludes anesthesia, or ASA Class 5
* EC18 Receiving anti-angiogenic treatment
* EC19 History of any coronary revascularization within the previous one (1) month.
* EC20 History of a stroke within the previous six (6) months.
* EC21 Anticipated need for any immunosuppressive drugs (including glucocorticoids).
* EC22 Subjects with severe non-proliferative or proliferative retinopathy.
* EC23 Patients with active known alcohol or illicit drug abuse.
* EC24 Severe comorbidity (i.e. cardiac or pulmonary) or poor general physical/mental health that, in the opinion of the Investigator, will not allow the subject to be a suitable study candidate (i.e. other advanced disease processes, diminished mental capacity, substance abuse, shortened life expectancy (≤1 year), etc.).
* EC25 The patient is currently involved in another clinical study.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Major Limb Amputation Free Survival | 12 months
  The measure of survival without a major (above the ankle) amputation within 12 months from the procedure and between group analyses at 12 months.

SECONDARY OUTCOMES:
Major amputation | 12 months
  Above the ankle amputation
All-Cause Mortality | 12 months
  Death from any cause
Doubling of wound size | 12 months
  Proportion of wounds that have doubled in size (area)
New full thickness lesion | 12 months
  New full thickness lesion (>1 cm2) on the index limb.
Wound healing (photographic method of measuring area, depth, perimeter and volume of wounds) | 1, 3, 6 and 12 months
  Quantitative evaluation of wound area continuous metric data (sq.cm.)
Wound healing (photographic method of measuring area, depth, perimeter and volume of wounds) | 1, 3, 6 and 12 months
  Quantitative evaluation of wound depth and perimeter in continuous metric data (cm)
Wound healing (photographic method of measuring area, depth, perimeter and volume of wounds) | 1, 3, 6 and 12 months
  Quantitative evaluation of wound volume in continuous metric data (cu.cm.)
Quality of Life Assessment (a PAD-specific health-related quality of life instrument) | 1, 3, 6, and 12 months
  VascuQoL Questionnaire (using subjective, ordinal data regarding patient life style on a scale of 1-7, where 1="all of the time", and 7= "none of the time").
Quality of Life Assessment (a PAD-specific health-related quality of life instrument) | 1, 3, 6, and 12 months
  VascuQoL Questionnaire (using subjective, ordinal data regarding patient discomfort on a scale of 1-7, where 1="A very great deal of discomfort or distress", and 7= "no discomfort or distress").
Quality of Life Assessment (a PAD-specific health-related quality of life instrument) | 1, 3, 6, and 12 months
  VascuQoL Questionnaire (using subjective, ordinal data regarding activity on a scale of 1-7, where 1="Totally limited, couldn't go shopping at all", and 7= "not at all limited").
Quality of Life Assessment (a PAD-specific health-related quality of life instrument) | 1, 3, 6, and 12 months
  VascuQoL Questionnaire (using subjective, ordinal data regarding walking improvement on a scale of 1-7, where 1="Not at all", and 7= "a very great deal").
Skin Perfusion Pressure (SPP) | 1, 3, 6 and 12 months
  Limb pressure measurement as a proxy for tissue perfusion

OTHER OUTCOMES:
Ankle Brachial Index (ABI) | 1, 3, 6 and 12 months
  Also a proxy for limb perfusion
Rest Pain | 1, 3, 6 and 12 months
  Rest Pain assessment using visual analog scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Dalip Sethi, PhD, Study Director — Cesca Therapeutics, Inc.